CLINICAL TRIAL: NCT06601920
Title: A Study of Activity Leader to Forest Therapy Campaign in Different Environments Targets on the Participants Which Had Been Infected by SARS-COV-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: Forestry Research Institute, Ministry of Agriculture, Taiwan (Unknown)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Superintendent, Branch of Linsen Chinese Medicine and Kunming, Taipei City Hospital, Taipei City Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TCHIRB-11112011; 112A040-04 (Other Grant/Funding Number: Forestry Research Institute, Ministry of Agriculture, Taiwan)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post COVID-19 Syndrome; Stress Disorders; Life Quality; Depression Anxiety Disorder
Keywords: Post COVID-19 syndrome; Profile of Mood States 2nd Edition-Adult Short,POMS; The Beck Depression In- ventory-Second edition, BDI-II; The Beck Anxiety Inventory, BAI; WHOQOL-BREF
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Stress Disorders, Traumatic | interventions — Forest Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Guided and then self-guided in Taipei Botanical Garden (Experimental): One group will get guided forest healing activities during the first period of the trial, and then self-guided during the second period in Taipei Botanical Garden.
  Interventions: Behavioral: Forest healing activities
- Self-guided and then guided in Taipei Botanical Garden (Experimental): One group will get "self-guided healing activities" during the first period of the trial, and then "guided forest healing activities" during the second period in Taipei Botanical Garden.
  Interventions: Behavioral: Forest healing activities
- Guided and then self-guided in Chiayi Arboretum. (Experimental): One group will get "guided forest healing activities" during the first period of the trial, and then "self-guided healing activities" during the second period in Chiayi Arboretum.
  Interventions: Behavioral: Forest healing activities
- Self-guided and then guided in Chiayi Arboretum (Experimental): One group will get "self-guided healing activities" during the first period of the trial, and then "guided forest healing activities" during the second period in Chiayi Arboretum.
  Interventions: Behavioral: Forest healing activities

INTERVENTIONS:
Behavioral: Forest healing activities — The two-hour forest healing activity, led by horticultural therapists from the Taiwan Horticultural Therapy Association, includes activities such as leaf stacking on stones, listening to sounds with closed eyes, body stretching, blindfolded tree identification, "my tree friend," earth mandala creation, tea tasting, and sharing of reflections.
  Other Names: Forest therapy

SUMMARY:
The goal of this clinical trial is to investigate the impact of self-guided forest healing activities and guided forest healing activities on the reduction of psychological stress inindividuals diagnosed with the new coronavirus. The main questions aim to answer are:

1. Effectiveness of Forest Healing Activities on Emotional Well-being: Researchers will compare the emotional improvement effects between self-guided and guided forest healing activities to determine their effectiveness.
2. Comparison of Healing Effects in Different Locations: Researchers will compare the effects of forest healing activities conducted in two similar environments, the Taipei Botanical Garden and the Chiayi Arboretum, to assess whether location influences outcomes despite similar altitude and latitude.

Participants who have been diagnosed with the new coronavirus will be recived two hours of guided forest healing activities or self-guided forest healing activities.

DETAILED DESCRIPTION:
In response to the psychosocial conditions arising from the ongoing pandemic, forest healing offers a corresponding solution. Forest healing activities have shown good adaptability in addressing conditions such as depression and anxiety. A systematic big data analysis paper highlights a significant decrease in depression following forest healing, with a Test overall effect Z=-6.204, as well as a similar significant reduction in anxiety with a Test overall effect Z=-4.183 (Yeon et al., 2021). For urban dwellers, a systematic review of big data on healing activities conducted in forest environments demonstrates significant normalization of systolic and diastolic blood pressure, an increase in the parasympathetic-to-sympathetic nervous system ratio, and a reduction in salivary cortisol concentration, with blood pressure shifting closer to normal indicators and salivary cortisol levels showing a downward trend after activities (Park et al., 2010; Qiu et al., 2022). Among populations exposed to chronic stressors, cortisol levels are higher compared to normal groups (Miller et al., 2007), and elevated salivary amylase activity is also noted compared to control groups (Vineetha et al., 2014). Therefore, forest healing significantly improves conditions like anxiety and depression, as reflected in the reduction of salivary cortisol concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been diagnosed with COVID-19 (SARS-CoV-2) and have completed their isolation.
* Participants aged 18 years or older who voluntarily agree to participate in the study.

Exclusion Criteria:

* Individuals who do not have the capability and stamina to walk for more than 120 minutes.
* Current smokers, betel nut chewers, or individuals who consume alcohol (more than five standard drinks in any situation).
* Individuals with a history of substance addiction (including both narcotic and non-narcotic drugs).
* Participants currently involved in another clinical trial or undergoing an intervention trial follow-up.
* Pregnant or breastfeeding women.
* Situations where participants are unable to cooperate (e.g., inability to participate after random assignment or refusal to sign the informed consent form).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States 2nd Edition-Adult Short, POMS | Before and after the two-hour forest healing activity
  The POMS (Profile of Mood States) is an indicator of both negative and positive emotions. It is divided into measures of positive social interaction (Friendliness), positive emotion scores, and negative emotion scores. A higher total POMS mood disturbance score (POMSTMD) indicates that negative emotions outweigh positive ones, while a lower score indicates the opposite.
  POMS contains 35 emotional adjectives, and participants select the option that best describes their emotional state for each adjective. The response options are: not at all, moderately, and extremely, scored from 0 to 4, respectively.
  The total score is calculated by subtracting the positive emotion Vigor score from the sum of the negative emotion subscale scores. Subscale scores range from 0 to 20, and the total score ranges from -20 to 100, with a minimum scale difference of 1 point.
The Beck Anxiety Inventory, BAI | Before the two-hour forest healing activity and again 7 days afterward.
  The BAI (Beck Anxiety Inventory) is a self-assessed anxiety scale developed by the research team at the Center for Cognitive Therapy, Department of Psychiatry, University of Pennsylvania School of Medicine. It asks participants to rate their level of distress for 21 anxiety-related symptoms. The response options are: not at all, mildly, moderately, and severely, with scores ranging from 0 to 3.
  The scale consists of 21 items, with each item scored from 0 to 3. The total score ranges from 0 to 63, with a minimum scale difference of 1 point. Scores of 0-7 indicate minimal anxiety, 8-15 indicate mild anxiety, 16-25 indicate moderate anxiety, and 26-63 indicate severe anxiety.
The Beck Depression In- ventory-Second edition, BDI-II | Before the two-hour forest healing activity and again 14 days afterward.
  The BAI (Beck Anxiety Inventory) is a self-assessed anxiety scale developed by the research team at the Center for Cognitive Therapy, Department of Psychiatry, University of Pennsylvania School of Medicine. It asks participants to rate their level of distress for 21 anxiety-related symptoms. The response options are: not at all, mildly, moderately, and severely, with scores ranging from 0 to 3.
  The scale consists of 21 items, with each item scored from 0 to 3. The total score ranges from 0 to 63, with a minimum scale difference of 1 point. Scores of 0-7 indicate minimal anxiety, 8-15 indicate mild anxiety, 16-25 indicate moderate anxiety, and 26-63 indicate severe anxiety.
The brief World Health Organization Quality of Life, WHOQOL-BREF | Before the two-hour forest healing activity and again 28 days afterward.
  The WHOQOL-BREF is the abbreviated version of the World Health Organization Quality of Life Questionnaire (WHOQOL-100), which defines quality of life as an individual's perception of their position in life within the context of the cultural value systems in which they live. This perception is related to six main areas: physical health, psychological state, level of independence, social relationships, personal beliefs, and environment. These are broken down into 24 facets, with each facet represented by one question. Additionally, two Taiwan-specific questions are included, forming the Taiwan abbreviated version of the questionnaire, which measures overall quality of life.
  The scale consists of 28 items, with higher scores indicating better quality of life. Each item is originally scored on a scale from 0 to 1, with a total score range of 0 to 28, and the minimum scale difference being 0.25 points.
Fear of COVID-19 Scale, FCV-19S | Before the two-hour forest healing activity and again 28 days afterward.
  The FSV-19S consists of 7 items, measuring participants' self-assessed fear of COVID-19. The results capture aspects of fearful thoughts, physiological reactions, and basic fears. The scale was reduced from 10 items to 7, with the items showing high intercorrelation. Responses are rated on a 5-point scale, ranging from strongly disagree, disagree, uncertain, agree, to strongly agree, scored from 1 to 5.
  The scale consists of 7 items, with each item scored from 1 to 5. The total score ranges from 7 to 35, with a minimum scale difference of 1 point.
Salivary Amylase Enzyme Activity | Before and after the two-hour forest healing activity
  Participants are required to collect saliva samples in microcentrifuge tubes with a capacity of at least 0.5 to 1.5 milliliters.
  Salivary Amylase Enzyme Activity Measurement: This is conducted using the SALIMETRICS® SALIVARY α-AMYLASE KINETIC ENZYME ASSAY KIT (Item No. 1-1902). The kit utilizes a compound formed by the covalent bonding of 2-chloro-p-nitrophenol and maltotriose, which is first hydrolyzed in a 96-well plate to produce maltotriose and 2-chloro-p-nitrophenol. The α-amylase in the saliva sample then converts 2-chloro-4-nitrophenylmaltoside into a product with an absorbance peak at 405 nm. The rate of this conversion determines the α-amylase activity.
Salivary Cortisol Concentration | Before and after the two-hour forest healing activity
  Participants are required to collect saliva samples in microcentrifuge tubes with a capacity of at least 0.5 to 1.5 milliliters.
  Salivary Cortisol Concentration Measurement: This is performed using the SALIMETRICS® Expanded Range High Sensitivity SALIVARY CORTISOL ENZYME IMMUNOASSAY KIT (Item No. 1-3002). The assay involves an enzyme-linked immunoassay with a four-parameter logistic model for calculation. Absorbance is read at a wavelength of 450 nm, with 490-492 nm used as a two-point calibration range. A higher reading corresponds to a lower concentration. The Salimetrics® kit includes a complete set of standards to minimize preparation errors.

SECONDARY OUTCOMES:
Post-COVID Functional Status, PCFS | Before the two-hour forest healing activity and again 28 days afterward.
  The PCFS (Post-COVID Functional Status) is a single-item functional assessment scale used to evaluate the impact on daily life following a COVID-19 diagnosis. The scale consists of only one question, with scores ranging from 0 to 4, and a minimum scale difference of 1 point.
Blood pressure, Heart rate, and Heart rate variability | Before and after the two-hour forest healing activity
  ANSWatch TS-0411 Heart Rate Master Wrist Physiological Monitor: This objective assessment tool measures indicators such as blood pressure, heart rate, and heart rate variability (HRV), providing insights into the participant's autonomic nervous system stability. The Heart Rate Master Wrist Physiological Monitor is a non-invasive, wearable electronic device. It is worn on the wrist and automatically takes measurements once powered on. The participant should sit or lie down, and the measurement process takes approximately 6-7 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, MD., PhD., Study Chair — Branch of Linsen Chinese Medicine and Kunming, Taipei City Hospital
Locations (1):
- Branch of Linsen Chinese Medicine and Kunming, Taipei City Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We undecided to share individual participant data (IPD) from this study. This decision is based on several factors:
  1. Privacy and Confidentiality: Protecting participant privacy is a priority, and sharing IPD could potentially compromise confidentiality despite de-identification efforts.
  2. Consent Limitations: The consent obtained from participants does not include provisions for sharing their individual data. We have not sought additional consent for data sharing.
  3. Data Security: Ensuring the security of sensitive personal data is challenging, and we do not have the resources to implement the necessary measures for secure data sharing.
  While we acknowledge the potential benefits of IPD sharing for advancing research, these considerations necessitate our current decision. We remain committed to adhering to ethical standards and protecting participant privacy.

REFERENCES:
- [Background] Yue Y, Li L, Liu R, Zhang Y, Zhang S, Sang H, Tang M, Zou T, Shah SM, Shen X, Chen J, Wu A, Jiang W, Yuan Y. The dynamic changes of psychosomatic symptoms in three waves of COVID-19 outbreak and fatigue caused by enduring pandemic in China. J Affect Disord. 2023 Jun 15;331:17-24. doi: 10.1016/j.jad.2023.03.032. Epub 2023 Mar 18. PMID 36934851
- [Background] Yeon PS, Jeon JY, Jung MS, Min GM, Kim GY, Han KM, Shin MJ, Jo SH, Kim JG, Shin WS. Effect of Forest Therapy on Depression and Anxiety: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Dec 1;18(23):12685. doi: 10.3390/ijerph182312685. PMID 34886407
- [Background] Voitsidis P, Nikopoulou VA, Holeva V, Parlapani E, Sereslis K, Tsipropoulou V, Karamouzi P, Giazkoulidou A, Tsopaneli N, Diakogiannis I. The mediating role of fear of COVID-19 in the relationship between intolerance of uncertainty and depression. Psychol Psychother. 2021 Sep;94(3):884-893. doi: 10.1111/papt.12315. Epub 2020 Nov 20. PMID 33216444
- [Background] Vineetha R, Pai KM, Vengal M, Gopalakrishna K, Narayanakurup D. Usefulness of salivary alpha amylase as a biomarker of chronic stress and stress related oral mucosal changes - a pilot study. J Clin Exp Dent. 2014 Apr 1;6(2):e132-7. doi: 10.4317/jced.51355. eCollection 2014 Apr. PMID 24790712
- [Background] Qiu Q, Yang L, He M, Gao W, Mar H, Li J, Wang G. The Effects of Forest Therapy on the Blood Pressure and Salivary Cortisol Levels of Urban Residents: A Meta-Analysis. Int J Environ Res Public Health. 2022 Dec 27;20(1):458. doi: 10.3390/ijerph20010458. PMID 36612777
- [Background] Park BJ, Tsunetsugu Y, Kasetani T, Kagawa T, Miyazaki Y. The physiological effects of Shinrin-yoku (taking in the forest atmosphere or forest bathing): evidence from field experiments in 24 forests across Japan. Environ Health Prev Med. 2010 Jan;15(1):18-26. doi: 10.1007/s12199-009-0086-9. PMID 19568835
- [Background] Lam ICH, Wong CKH, Zhang R, Chui CSL, Lai FTT, Li X, Chan EWY, Luo H, Zhang Q, Man KKC, Cheung BMY, Tang SCW, Lau CS, Wan EYF, Wong ICK. Long-term post-acute sequelae of COVID-19 infection: a retrospective, multi-database cohort study in Hong Kong and the UK. EClinicalMedicine. 2023 Jun;60:102000. doi: 10.1016/j.eclinm.2023.102000. Epub 2023 May 11. PMID 37197226
- [Background] Labrague LJ, de Los Santos JAA. Fear of COVID-19, psychological distress, work satisfaction and turnover intention among frontline nurses. J Nurs Manag. 2021 Apr;29(3):395-403. doi: 10.1111/jonm.13168. Epub 2020 Oct 11. PMID 32985046
- [Background] Kim JG, Shin WS. Forest Therapy Alone or with a Guide: Is There a Difference between Self-Guided Forest Therapy and Guided Forest Therapy Programs? Int J Environ Res Public Health. 2021 Jun 29;18(13):6957. doi: 10.3390/ijerph18136957. PMID 34209647
- [Background] Han Q, Zheng B, Agostini M, Belanger JJ, Gutzkow B, Kreienkamp J, Reitsema AM, van Breen JA, Collaboration P, Leander NP. Associations of risk perception of COVID-19 with emotion and mental health during the pandemic. J Affect Disord. 2021 Apr 1;284:247-255. doi: 10.1016/j.jad.2021.01.049. Epub 2021 Jan 26. PMID 33602537
- [Background] Dye C. Health and urban living. Science. 2008 Feb 8;319(5864):766-9. doi: 10.1126/science.1150198. PMID 18258905